CLINICAL TRIAL: NCT06328088
Title: Effect of Vegetarian Versus Non Vegetarian Based Diet in the Recurrence of Hepatic Encephalopathy in Patients With Cirrhosis:An Open Label Study
Brief Title: Vegetarian Versus Non Vegetarian Based Diet in the Recurrence of Hepatic Encephalopathy in Patients With Cirrhosis: An Open Label Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr. Praveen Shrama, Professor, Sir Ganga Ram Hospital
Other Study IDs: EC/12/23/2400
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic encephalopathy;diet;vegetarian;non vegetarian;cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non vegetarian diet: Non vegetarian diet
  Interventions: Dietary Supplement: Non vegetarian
- Vegetarian diet: Vegetarian diet
  Interventions: Dietary Supplement: Non vegetarian

INTERVENTIONS:
Dietary Supplement: Non vegetarian — Non vegetarian diet plus supportive treatment including lactulose and/or rifaximin

SUMMARY:
Earlier protein restriction was advocated in the treatment of HE but later this concept was refuted and increase protein intake was advocated in patients with HE. Diet in patients during an episode HE is also not known. It is advisable based on many case reports or case series that vegetable-based diet during the episode of HE is better than animal-based diet as it reduces ammonia level and other false neurotransmitters in brain and helps in early recovery of, HE . However, diet in patients who had recovered from an episode of, HE is not known and what type of protein (vegetarian or non-vegetarian) should be taken to prevent another episode of HE has never been evaluated. In India majority of the patients are vegetarian and patients with cirrhosis are malnourished and lack protein in their diet as per our previous published study

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a neurological complication in cirrhosis and affects 30-80% of these patients. Patient conscious level varies from minimal altered sensorium to deep coma and hence it is classified into two categories, covert HE and overt HE. Its occurrence in patients with cirrhosis merits liver transplantation and it reduces survival rate to 50% in next 1-2 year. HE significantly affects quality of life, inability to drive, morbidity and mortality . Recovery from single episode of HE merits secondary prophylaxis with lactulose and rifaximin .

Protein calorie malnutrition is also common in patients with cirrhosis and its prevalence varies from 30-90% depending upon the method of evaluation and types of patients enrolled . Sarcopenia negatively affects survival and can be precipitated by repeated episodes of admission and HE in patients with cirrhosis. Earlier protein restriction was advocated in the treatment of HE but later this concept was refuted and increase protein intake was advocated in patients with HE . Diet in patients during an episode HE is also not known. It is advisable based on many case reports or case series that vegetable-based diet during the episode of HE is better than animal-based diet as it reduces ammonia level and other false neurotransmitters in brain and helps in early recovery of, HE . However, diet in patients who had recovered from an episode of, HE is not known and what type of protein (vegetarian or non-vegetarian) should be taken to prevent another episode of HE has never been evaluated. In India majority of the patients are vegetarian and patients with cirrhosis are malnourished and lack protein in their diet as per our previous published study . We wish to study effect of diet on the recurrence of HE in patient with cirrhosis who had recovered completely from an episode of HE and are on secondary prophylaxis of HE.

Materials and methods:

Consecutive patients with cirrhosis who have recovered from an episode of HE will be screened and enrolled in the study if fulfilling the enrolment criteria. Cirrhosis will be diagnosed based on clinical, radiological, Transient elastography and biopsy if available. All relevant investigation will be done to evaluate the cause of cirrhosis (Viral markers, autoimmune markers etc). HE will be diagnosed based on West Heaven criteria and recovery will be assessed by the senior Consultant of this study. All patient will undergo handgrip strength test to assess muscle strength, number connection test and critical flicker frequency test to assess minimal hepatic encephalopathy at baseline and at 1,3 and 6 month interval.

Handgrip test: This is a simple bed side test non-invasive tests in which patient will sit on a chair and held a instrument and press it as hard as possible after a training session to get the muscle strength. Its value will be recorded (26).

Number connection test: It is simple bed side paper and pencil tests.In a paper numbers are written from 1 to 25 in a random session and patient will join the number as fast as possible and result will be recorded(4) Critical flicker frequency tests: It is again a simple bed side test in which patient will see an instrument and a light source. Patient will see the flickering of light and he will record it by pushing a button. Its value will be recorded(27).

Blood tests which includes complete blood count,liver and kidney function tests,INR will be assessed at baseline,1,3 and 6 month as per standard practise in these patients.

Assessment of dietary intake All patients will be assessed by investigator and trained dietician for the calculation of total calories, carbohydrates, protein and fat by 24 recall method. Assessment of these parameters will be compared as per standard recommendation by INASL guidelines(10). If patient is taking less calories or proteins, these will be supplemented according to patient choice of food and as per standard guidelines.

Vegetarian subjects: Protein will be supplemented as per recommendation 1.5 gm/kg body weight and it will be supplemented with vegetable source. Milk and milk products are allowed in this group as most of the Indians who are vegetarian also consume milk and milk products. Egg and meat products are not allowed.

Non vegetarian subjects: Protein will be supplemented by both vegetarian and non-vegetarian diet. Patients will be encouraged to take more>50% of total daily protein requirement as non-vegetarian based protein which will include eggs and meat products. Due to cultural belief in India people do not take non vegetarian food on daily basis. Patients will maintain a dairy of their daily protein source. If patient is taking less than 50% of his daily protein from non-vegetarian source for more than 10 days per month these patients will be taken as non-compliant and will be recorded.

Randomisation protocol: This will be an open label study and patients will be divided into two groups based on their dietary pattern previous to enrolling in this study. Patients who are strict vegetarian will be grouped into vegetarian group and patients who are non vegetarian will be given a choice to enrol in any group and will be randomised accordingly.

Follow up protocol:

All patients will be followed by the investigator at baseline, fifteen days and then at one month interval for 6 months from day of enrolment in the study. All patients are free to come to hospital at any time in case of any medical issue and will be assessed as per standard protocol. All patients will be managed as per standard practise and all previous medications like beta blockers, diuretics, antiviral therapy, lactulose and rifaximin will be continued if taking. Patient on secondary prophylaxis for HE with lactulose with or without rifaximin will continue the medications.

Management of Hepatic encephalopathy: All patients will be managed as per standard protocol with correction of precipitating factors, lactulose, L ornithine L aspartate infusion or sachets and rifaximin. Patients with more than grade 2 encephalopathy will be admitted

Statistical methods:

The results of this study will be expressed as mean± standard error. The p value of < 0.05 will be considered statistically significant. Data will be compared using the non-parametric Mann-Whitney test for continuous data and Fisher test for categorical data. Comparisons of the variables will be performed using the Wilcoxon test and Fisher test as needed. Statistical analyses of the data will be performed by using SPSS 23 Statistical Software (SPSS Inc. and Microsoft Corp., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

- 1) Age 18 years and older. 2) Confirmed diagnosis of liver cirrhosis. (Diagnosed on the basis of clinical, biochemical, radiological or endoscopic features).

3) Willingness to sign informed consent proforma. 4) Patients who recovered from Hepatic encephalopathy will be enrolled from Out patient Department within 15 days of discharge

Exclusion Criteria:

- 1) Patients with underlying severe cardiopulmonary disease or hepatocellular carcinoma.

2) Patients with CTP score of more than 12 3) Patient not willing for follow up or consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of cirrhosis and hepatic encephalopathy who has completely recovered from Hepatic encephalopathy and put on secondary prophylaxis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Recurrence of overt hepatic encephalopathy | 6 month follow up

SECONDARY OUTCOMES:
Hospitalization due to any cause | six month

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital, Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided